CLINICAL TRIAL: NCT02069600
Title: OBSTRUCTIVE SLEEP APNEA IN THE ELDERLY. ROLE OF CONTINUOUS POSITIVE AIRWAY PRESSURE TREATMENT. A Randomized Controlled Trial
Brief Title: Effect of CPAP Treatment in Elderly: Randomized Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario La Fe (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Miguel Angel Martinez-Garcia, MD, PhD, Hospital Universitario La Fe
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT-elderly-OSA
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Elderly; CPAP; clinical trial; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Positive Airway Pressure (Active Comparator): Continuous Positive Airway Pressure is a device that apply a positive pressure in the airway to avoid its collapse during sleep during three months in this study
  Interventions: Device: Continuous Positive Airway Pressure
- No intervention (No Intervention): No intervention. No placebo is used. Control group without CPAP treatment during three months

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — CPAP applies a positive pressure into the airway to avoid its collapse during sleep.
  The pressure used in each patient is calculate by an auto CPAP device during 3 months. This device calculate the pressure that avoid 95% of sleep-disordered breathing
  Other Names: CPAP device from ResMed CO. Sydney.
  Arms: Continuous Positive Airway Pressure

SUMMARY:
Rationale: Almost all the information the investigators have about the effect of continuous positive airway pressure (CPAP) in patients with obstructive sleep apnea (OSA) comes from randomized clinical trials including only middle-aged patients. Little is know, however, about the effect of CPAP in elderly people with OSA. Objective: To assess the effect of CPAP treatment in elderly patients with severe OSA on clinical, quality-of-life and neurocognitive spheres. Methods and Measurements: Open-label, randomized, multicenter clinical trial of parallel groups with blinded end-point design conducted in 12 Spanish teaching hospitals on a consecutive clinical cohort of elderly (≥ 70 years) patients with confirmed severe OSA (IAH≥ 30) receiving CPAP or no therapy while maintaining their usual control for three months. CPAP titration was performed by an auto CPAP device. A good adherence was set as at least 4 hours/day of CPAP use. Primary endpoint was the measurement of quality of life by the Quebec Sleep questionnaire, which includes diurnal and nocturnal symptoms, hypersomnolence, and social and emotional dimensions. Secondary endpoints include different sleep-related symptoms, presence of anxiety or depression, office blood pressure figures and some neurocognitive tests. Patients were invited to a clinical visit on three occasions to quantify the adherence to CPAP. Intention-to-treat analysis was performed.

DETAILED DESCRIPTION:
Not needed

ELIGIBILITY:
Inclusion Criteria:

* Patients were initially eligible for participation in the study if they were aged at least 70 years, had an apnea-hypopnea index (AHI) ≥30 and had signed the informed consent to participate

Exclusion Criteria:

* Current use of CPAP treatment, central sleep apnea (defined as at least 50% of respiratory events having a pattern of apnea or hypopnea without respiratory effort), respiratory failure (defined as diurnal oxygen saturation below 90%), severe heart failure (NYHA III-IV), a cardiovascular event in the month prior to the inclusion in the study or disabling hypersomnia requiring urgent treatment (defined as an Epworth Sleepiness Scale ≥ 18).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 224 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Quality of life | Changes in quality baseline from baseline to 3 months after random
  Quality of life measure by Quebec Sleep Questionnaire (QSQ). This is an specific sleep questionnaire

SECONDARY OUTCOMES:
Sleep-related symptoms | Changes in sleep-related symptoms from baseline to three months after random
  Snoring Witnessed apnea Choking Hypersomnolence Nocturia Nightmares

OTHER OUTCOMES:
Neurocognitive tests | Changes in neurocognitive tests from baseline to three months after random
  Trail-Making-Test A Trail-Making-Test B Digital Symbol Test Digit Span Test Hospital Depression and Anxiety test Epworth test
Office Blood pressure measurements | Changes in blood pressure levels from baseline to three months after random
  3 office Systolic blood pressure and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Martinez Martínez García, MD, PhD, Principal Investigator — Hospital La Fe Valwncia
Locations (1):
- Hospital Universitario La Fe Valwncia, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Martinez-Garcia MA, Oscullo G, Ponce S, Pastor E, Orosa B, Catalan P, Martinez A, Hernandez L, Muriel A, Chiner E, Vigil L, Carmona C, Mayos M, Garcia-Ortega A, Gomez-Olivas JD, Beauperthuy T, Bekki A, Gozal D. Effect of continuous positive airway pressure in very elderly with moderate-to-severe obstructive sleep apnea pooled results from two multicenter randomized controlled trials. Sleep Med. 2022 Jan;89:71-77. doi: 10.1016/j.sleep.2021.11.009. Epub 2021 Nov 24. PMID 34915264
- [Derived] Martinez-Garcia MA, Chiner E, Hernandez L, Cortes JP, Catalan P, Ponce S, Diaz JR, Pastor E, Vigil L, Carmona C, Montserrat JM, Aizpuru F, Lloberes P, Mayos M, Selma MJ, Cifuentes JF, Munoz A; Spanish Sleep Network. Obstructive sleep apnoea in the elderly: role of continuous positive airway pressure treatment. Eur Respir J. 2015 Jul;46(1):142-51. doi: 10.1183/09031936.00064214. Epub 2015 May 28. PMID 26022945